CLINICAL TRIAL: NCT02373540
Title: Real-world Evaluation of Outcome Data Under a Prospective, Observational, Post-Market Clinical Study, Using the Algovita SCS System to Treat Patients With Chronic Pain of the Trunk and/or Limbs Per the Applicable Indications for Use
Brief Title: Algovita Post-Market Clinical Study: Spinal Cord Stimulation to Treat Chronic Pain
Status: Terminated | Type: Observational
Sponsor: Nuvectra (Industry)
Collaborators: Bright Research Partners (Industry)
Responsible Party: Sponsor
Other Study IDs: CLPR 0236
Record Dates: First submitted 2015-02-23; First posted 2015-02-27 (Estimated); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: Chronic Pain
Keywords: spinal cord stimulation; chronic pain; failed back surgery syndrome
MeSH Terms: conditions — Chronic Pain; Failed Back Surgery Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Algovita Spinal Cord Stimulation system

SUMMARY:
The purpose of this study is to obtain real-world clinical outcome data for the Algovita Spinal Cord Stimulation system when used, on-label, according to the applicable directions for use.

ELIGIBILITY:
Inclusion Criteria:

* Patient is eligible for SCS therapy according to the Algovita SCS system Indications for Use statement
* Patient had successful Algovita SCS system stimulation trial with an Algovita SCS system and will be implanted with a permanent Algovita SCS system; prior approval must be obtained from the Sponsor if another SCS system was used for the stimulation trial
* Patient is willing and able to sign an IRB/EC approved informed consent, and in the United States, a Privacy Protection Authorization, as required

Exclusion Criteria:

* Patient is contraindicated for an Algovita SCS system
* Patient has a cognitive impairment, or exhibits any characteristic, that would limit study candidate's ability to assess pain relief or complete study assessments
* Patient has a life expectancy of less than 2 years
* Patient is participating in another clinical study that would confound data analysis
* Patient has a coexisting pain condition that might confound pain ratings

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic, intractable pain of the trunk and/or limbs who are appropriate to receive SCS therapy and successfully complete a stimulation trial.
Sampling Method: Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Percent reduction in targeted pain compared to baseline | 6 Month Follow-up Visit
  Percentage of participants who experience at least a 50 percent reduction in targeted pain from baseline, as assessed by Numeric Rating Scale (NRS). The Numeric Rating Scale (NRS) will range from 0 to 10 with a higher score indicating a higher level of pain.

SECONDARY OUTCOMES:
Percent reduction in targeted pain compared to baseline | 1, 3, 12, 18, and 24 Month Follow-up Visits
  Percentage of participants who experience at least a 50 percent reduction in targeted pain from baseline, as assessed by Numeric Rating Scale (NRS). The Numeric Rating Scale (NRS) will range from 0 to 10 with a higher score indicating a higher level of pain.
Percent change in targeted pain intensity compared to baseline | 1, 3, 6, 12, 18, and 24 Month Follow-up Visits
  Percent reduction or actual reduction from baseline in targeted pain intensity, as assessed by Numeric Rating Scale (NRS). The Numeric Rating Scale (NRS) will range from 0 to 10 with a higher score indicating a higher level of pain.
Change in disability compared to baseline | 1, 3, 6, 12, 18, and 24 Month Follow-up Visits
  Change from baseline in disability as measured by Oswestry Disability Index (ODI). The Oswestry Disability Index is scored between 0 and 100 with higher scores indicating a greater disability.
Change in quality of life compared to baseline | 1, 3, 6, 12, 18, and 24 Month Follow-up Visits
  Change from baseline in quality of life as measured by EQ-5D, a standardized measure of health status.
Willingness to undergo procedure again | 1, 3, 6, 12, 18, and 24 Month Follow-up Visits
  To record the participants willingness to undergo the procedure again using a question (yes/no) if the participant would be willing to undergo the procedure again.
Rate of device-related and/or procedure-related Adverse Events (AEs) | From Implant through 24 Month Follow-up Visit
  To record the rate of device-related and/or procedure-related Adverse Events (AEs).
Rate of surgical intervention of the SCS system | From Implant through 24 Month Follow-up Visit
  To record the rate of surgical intervention of the SCS system.

CONTACTS AND LOCATIONS:
Overall Officials: Ben Tranchina, Study Director — Nuvectra
Locations (18):
- United States (16):
  - Summit Healthcare Pain Clinic Associates, Show Low, Arizona
  - Coastal Pain and Spinal Diagnostics, Carlsbad, California
  - Samaritan Center for Medical Research, Los Gatos, California
  - Restore Orthopedics and Spine Center, Orange, California
  - Vitamed Research, Rancho Mirage, California
  - Spine & Nerve Diagnostic Center, Roseville, California
  - Relieve Pain Center, San Diego, California
  - Nona Medical Arts, Orlando, Florida
  - South Florida Clinical Research, South Miami, Florida
  - Ephraim McDowell Regional Medical Center, Danville, Kentucky
  - Brigham and Women's Hospital, Chestnut Hill, Massachusetts
  - Nevada Advanced Pain Specialists, Reno, Nevada
  - Garden State Pain Control, Clifton, New Jersey
  - OMNI Pain and Precision Medicine, Utica, New York
  - St. Luke's University Health Network, Bethlehem, Pennsylvania
  - Pennsylvania Pain and Spine, Chalfont, Pennsylvania
- Germany (2):
  - Universitatksklinikum Dusseldorf, Düsseldorf
  - NCN-Neurochirurgische Praxis Neuss, Neuss